CLINICAL TRIAL: NCT06529822
Title: Phase 1 Clinical Trial of a Personalized Cancer Vaccine (PCV) Strategy in Patients With Solid Tumors and Molecular Residual Disease
Brief Title: Personalized Cancer Vaccine (PCV) Strategy in Patients With Solid Tumors and Molecular Residual Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202412028
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Muscle-Invasive Bladder Carcinoma; Gastroesophageal Adenocarcinoma
Keywords: Personalized cancer vaccine; Solid tumor; Immunotherapy; Bladder cancer; Gastroesophageal Adenocarcinoma; GEC
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Cohort 1: Muscle Invasive Bladder Cancer (PCV) (Experimental): The schedule for vaccination will be Days 1, 4, 8, 15, 29, 57, 85, 113, 141, and 169. All study injections will be given intramuscularly and co-administered with poly-ICLC by a trained healthcare provider.
  Interventions: Biological: Synthetic long peptide personalized cancer vaccine; Drug: Poly ICLC; Device: Signatera assay
- Cohort 2: Gastroesophageal Adenocarcinoma (GEC) (Experimental): The schedule for vaccination will be Days 1, 4, 8, 15, 29, 57, 85, 113, 141, and 169. All study injections will be given intramuscularly and co-administered with poly-ICLC by a trained healthcare provider.
  Interventions: Biological: Synthetic long peptide personalized cancer vaccine; Drug: Poly ICLC; Device: Signatera assay

INTERVENTIONS:
Biological: Synthetic long peptide personalized cancer vaccine — Neoantigen vaccines will be provided on a patient-specific basis
  Other Names: PCV
Drug: Poly ICLC — Poly-ICLC will be supplied by Oncovir, Inc.
  Other Names: Hiltonol
Device: Signatera assay — Signatera is a clinically validated, personalized, tumor-informed, multiplex-PCR and next-generation sequencing (NGS) based clinical trial assay targeting 16 tumor-specific mutations. It is intended for the detection of ctDNA isolated from anticoagulated peripheral whole blood from post-surgical patients previously diagnosed with localized or advanced solid tumors to aid physician assessment and treatment decision-making, together with other clinical factors

SUMMARY:
This is a phase 1 clinical trial to evaluate the safety, feasibility and immunogenicity of a personalized cancer vaccine strategy in patients with solid tumors and molecular residual disease. The hypothesis of the trial is that synthetic long peptide personalized cancer vaccines will be safe and capable of generating measurable neoantigen-specific T-cell responses enabling ctDNA clearance. The personalized cancer vaccines are composed of synthetic long peptides corresponding to prioritized cancer neoantigens and will be co-administered with poly-ICLC.

ELIGIBILITY:
Inclusion Criteria Cohort #1:

* Age ≥ 18 years.
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%).
* Histologically confirmed muscle-invasive bladder cancer (MIBC) or upper tract urothelial carcinoma (renal pelvis and/or ureter).
* Patients with carcinomas showing mixed histologies are required to have a dominant transitional cell pattern.
* Complete surgical resection of MIBC (R0) or upper tract urothelial carcinoma (renal pelvis and/or ureter). Tumor, nodes, metastases (TNM) classification (based on the American Joint Committee on Cancer (AJCC) Cancer Staging Manual 8th ed.) at pathological examination of surgical resection specimen as follows: pT2-4aN0M0 or pT0-4aN+M0.
* Patient must have fully recovered from surgical resection in the opinion of the treating MD.
* ctDNA positive result as identified by Signatera.
* Radiologic confirmation (by conventional imaging) of absence of residual disease and absence of metastasis.
* Adequate bone marrow and organ function as defined below:

  * WBC ≥ 1.5 K/cumm
  * Absolute neutrophil count ≥ 1.0 K/cumm
  * Platelets ≥ 50 K/cumm
  * Hemoglobin ≥ 8.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine clearance > 30 mL/min by Cockcroft-Gault
* The effects of synthetic long peptide personalized cancer vaccines and Hiltonol on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 5 months after completion of study interventions. Should a woman become pregnant or suspect she is pregnant while participating in this study or should a man suspect he has fathered a child, s/he must inform her treating physician immediately.
* No concurrent investigational therapies outside of this protocol are allowed.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria Cohort #1:

* Receiving any other investigational agents, or planning to receive other investigational agents as part of neoadjuvant therapy. Patients who have received perioperative neoadjuvant chemotherapy and immunotherapy are allowed.
* Known allergy, or history of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty.
* A psychiatric illness or social situations that would limit compliance with study requirements as determined by the investigator from the medical history, physical exam, and/or medical record.
* Prior or currently active autoimmune disease requiring management with immunosuppression. This includes inflammatory bowel disease, ulcerative colitis, Crohn's disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome, sarcoidosis, or other rheumatologic disease or any other medical condition or use of medication (e.g., corticosteroids) which might make it difficult for the patient to complete the full course of treatments or to generate an immune response to vaccines. In the case of asthma or chronic obstructive pulmonary disease taking inhaled corticosteroids that does not require daily systemic corticosteroids is acceptable. Additionally, local acting steroids (topical, inhaled, or intraarticular) will be allowed. Patients on intermittent or short course steroids will be allow if the dose does not exceed 4 mg of dexamethasone (or equivalent) per day for > 7 consecutive days. Premedication for chemotherapy does not apply to this criterion and may be administered as per SOC practice. Any patients receiving steroids should be discussed with the PI to determine if eligible.
* Pregnant and/or breastfeeding.
* Known HIV-positive status.
* History of positive test for Hepatitis B virus surface antigen (HBsAg) and/or positive Hepatitis C antibody result with detectable hepatitis C virus (HCV) ribonucleic acid (RNA) indicating acute or chronic infection
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia. For treatment enrollment the patient must have completed all prior cancer treatments > 28 days prior to vaccine administration with the exception of adjuvant SOC immunotherapy.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial per discussion with the PI.
* Currently receiving any other investigational agents.
* Live vaccine administered within 30 days prior to enrollment.
* Known allergy, or history of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty.
* Immunodeficiency, systemic steroid therapy, or any other immunosuppressive therapy within 30 days of enrollment.
* Active autoimmune disease (excluding diabetes mellitus and/or vitiligo), solid organ or allogeneic bone marrow transplant, or other known contraindications to receiving immunotherapy.
* Severe hypersensitivity (grade ≥ 3) to checkpoint inhibitors and/or any of its excipients.
* A psychiatric illness or social situations that would limit compliance with study requirements, as determined by the investigator from the medical history, physical exam, and/or medical record.
* Current pneumonitis, a history of (non-infectious) pneumonitis requiring steroids, or history of clinically significant interstitial lung disease.
* Active tuberculosis test within 3 months prior to treatment initiation.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum/urine pregnancy test within 7 days of study entry.

Inclusion Criteria Cohort #2:

* Age ≥ 18 years.
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%)
* Histologically confirmed gastroesophageal adenocarcinoma
* Stage II or III gastroesophageal adenocarcinoma (GEC).
* Complete surgical resection of GEC (R0). Full recovery from surgery and enrollment within 52 weeks following surgery with curative intent. Tumor, nodes, metastases (TNM) classification (based on the American Joint Committee on Cancer (AJCC) Cancer Staging Manual 8th ed.) at pathological examination of surgical resection specimen as follows:

  * Esophageal and Esophagogastric junction adenocarcinoma T1 N1-3 M0 or T2-4 N0-2M0.
  * Gastric adenocarcinoma T1-2 N1-3 M0 or T3-4 N0-3 M0.
* Patient must have fully recovered from surgical resection in the opinion of the treating MD.
* ctDNA positive result as identified by Signatera.
* Radiologic confirmation (by conventional imaging) of absence of residual disease and absence of metastasis.
* Adequate bone marrow and organ function as defined below:

  * WBC ≥ 1.5 K/cumm
  * Absolute neutrophil count ≥ 1.0 K/cumm
  * Platelets ≥ 50 K/cumm
  * Hemoglobin ≥ 8.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine clearance > 30 mL/min by Cockcroft-Gault
* The effects of synthetic long peptide personalized cancer vaccines and Hiltonol and on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 5 months after completion of study interventions. Should a woman become pregnant or suspect she is pregnant while participating in this study or should a man suspect he has fathered a child, s/he must inform her treating physician immediately.
* No concurrent investigational therapies outside of this protocol are allowed.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria Cohort #2:

* Receiving any other investigational agents or planning to receive other investigational agents as part of neoadjuvant therapy. Patients who have received perioperative neoadjuvant chemotherapy and immunotherapy are allowed.
* Known allergy, or history of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty.
* A psychiatric illness or social situations that would limit compliance with study requirements as determined by the investigator from the medical history, physical exam, and/or medical record.
* Prior or currently active autoimmune disease requiring management with immunosuppression. This includes inflammatory bowel disease, ulcerative colitis, Crohn's disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome, sarcoidosis, or other rheumatologic disease or any other medical condition or use of medication (e.g., corticosteroids) which might make it difficult for the patient to complete the full course of treatments or to generate an immune response to vaccines. In the case of asthma or chronic obstructive pulmonary disease taking inhaled corticosteroids that does not require daily systemic corticosteroids is acceptable. Additionally, local acting steroids (topical, inhaled, or intraarticular) will be allowed. Patients on intermittent or short course steroids will be allow if the dose does not exceed 4 mg of dexamethasone (or equivalent) per day for > 7 consecutive days. Premedication for chemotherapy does not apply to this criterion and may be administered as per SOC practice. Any patients receiving steroids should be discussed with the PI to determine if eligible.
* Pregnant and/or breastfeeding.
* Known HIV-positive status.
* History of positive test for Hepatitis B virus surface antigen (HBsAg) and/or positive Hepatitis C antibody result with detectable hepatitis C virus (HCV) ribonucleic acid (RNA) indicating acute or chronic infection.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia. For treatment enrollment the patient must have completed all prior cancer treatments > 28 days prior to vaccine administration with the exception of adjuvant SOC immunotherapy.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial per discussion with the PI.
* Currently receiving any other investigational agents.
* Live vaccine administered within 30 days prior to enrollment.
* Known allergy, or history of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty.
* Immunodeficiency, systemic steroid therapy, or any other immunosuppressive therapy within 30 days of enrollment.
* Active autoimmune disease (excluding diabetes mellitus and/or vitiligo), solid organ or allogeneic bone marrow transplant, or other known contraindications to receiving immunotherapy.
* Severe hypersensitivity (grade ≥ 3) to checkpoint inhibitors and/or any of its excipients.
* A psychiatric illness or social situations that would limit compliance with study requirements, as determined by the investigator from the medical history, physical exam, and/or medical record.
* Current pneumonitis, a history of (non-infectious) pneumonitis requiring steroids, or history of clinically significant interstitial lung disease.
* Active tuberculosis test within 3 months prior to treatment initiation.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum/urine pregnancy test within 14 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2033-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by treatment-emergent adverse events (TEAEs) | From 1st vaccine dose through 30 days following last dose of vaccine (estimated to be 13 months)
Safety as measured by treatment-related adverse events (TRAEs) | From 1st vaccine dose through 30 days following last dose of vaccine (estimated to be 13 months)
  -At least possibly related to vaccine therapy
Safety as measured by serious adverse events (SAEs) | From 1st vaccine dose through 30 days following last dose of vaccine (estimated to be 13 months)
  As defined in 21 CFR 312.32:
  Definition: an adverse event is considered "serious" if, in the view of the investigator, it results in any of the following outcomes:
  * Death
  * A life-threatening adverse event
  * Inpatient hospitalization or prolongation of existing hospitalization
  * A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * A congenital anomaly/birth defect
  * Any other important medical event that does not fit the criteria above but, based upon appropriate medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above
Feasibility as measured by the success of enrolling patients with molecular residual disease | Through 30 months
  The trial will be feasible if 8 patients with molecular residual disease are enrolled in 30 months
Feasibility as measured by the expected time frame for vaccine creation | Through 24 weeks
  The trial will be feasible if the vaccine is created within 24 weeks from signing of treatment consent to vaccine availability.
Feasibility as measured by the rate of successful vaccine delivery | Through 1st vaccine dose (estimated to be 24 weeks)
  The trial will be feasible if at least 50% of patients receive the vaccine

SECONDARY OUTCOMES:
Immune response as measured by ELISPOT analysis | Through 2 years after completion of treatment (estimated to be 2.5 years)
  Treatment screening, day 1, day 15, day 29, day 57, day 85, day 113, day 141, day 169, 1 year (optional), and 2 years (optional)
Molecular residual disease as evaluated by ctDNA clearance using the Signatera assay | Through completion of follow-up (estimated to be 66 months)
  Treatment screening, day 1, day 8, day 15, day 29, day 57, day 85, day 113, day 141, day 169, and during follow-up.
Recurrence-free survival (RFS) | Through completion of follow-up (estimated to be 66 months)
  Recurrence-free survival is defined as the rate of recurrence from treatment enrollment until disease recurrence per standard of care assessments, or until patient is off study, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: William Gillanders, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu